CLINICAL TRIAL: NCT01605981
Title: A Phase II, Non Randomized, Open Label, Trial Evaluating Nilotinib as Treatment for Newly Diagnosed CML Patients in Accelerated Phase.
Brief Title: Trial Evaluating Nilotinib as Treatment for Newly Diagnosed CML Patients in Accelerated Phase.
Acronym: MACS1881
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107EBR06
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2014-06

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: Nilotinib; CML patients; accelerated phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib oral (Experimental): Nilotinib oral dose of 400 mg BID (800 mg/day) continuous dosing for up to 24 months. Nilotinib oral dose of 300 mg BID (600 mg/day) continuous dosing in case of intolerance. Nilotinib oral dose of 400 mg QD (400 mg/day) continuous dosing in case of intolerance
  Interventions: Drug: AMN107

INTERVENTIONS:
Drug: AMN107

SUMMARY:
This is an open label, non randomized, prospective, multicenter, phase II clinical trial evaluating nilotinib 400 mg BID for the treatment of newly diagnosed CML-AP patients.

Patients enrolled into the study will receive 400mg of nilotinib, orally, twice daily (800mg/day)

DETAILED DESCRIPTION:
Patients will be evaluated for safety throughout the study and for response every month for the first 3 months, then every 3 months thereafter up to month 24.

BCR-ABL transcripts measurement by QRT-PCR and mutation analyses will be done on peripheral blood samples and cytogenetic analyses on bone marrow aspirates.

Laboratory tests (hematology, blood chemistry), ECG and physical examination will be done on every visit.

Drug pharmacokinetics will be assessed in this study. For the screening Baseline periods, see chart attached

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age > 18 years old;
* Diagnosis of Chronic Myeloid leukemia in Accelerated Phase (CML-AP);
* Patients with CML-AP(See Appendix 1) within 3 months of diagnosis (date of initial diagnosis is the date of first reported cytogenetic analysis). Standard conventional cytogenetic analysis must be done on bone marrow. FISH cannot be used for purpose of inclusion;
* Patients with atypical BCR-ABL transcripts are eligible (transcripts other then b2a2 an b3a2);
* No previous treatment with any antileukemic drugs with the exception of hydroxyurea (HU) and/or anagrelide. In emergent cases where the patient requires disease management while awaiting study start, commercial supplies of Gleevec/Glivec at any dose may be prescribed to the patient but for no longer than 2 weeks in duration;
* ECOG 0,1 or 2;
* Normal serum levels > LLN (lower limit of normal) or corrected to within normal limits with supplements, prior to the first dose of study medication, of potassium magnesium and calcium;
* AST and ALT < 2.5 x ULN (upper limit of normal) or < 5.0 x ULN if considered due to leukemia;
* Alkaline phosphatase < 2.5 x ULN, unless considered due to leukemia;
* Total bilirubin < 1.5 x ULN;
* Serum lipase and amylase < 1.5 x ULN;
* Written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Patients in Chronic and Blastic Phases.
* Patients who are considered Ph negative because they do not have a confirmed cytogenetic diagnosis of Philadelphia Ph+ chromosome (9;22 translocation) in > 20 metaphases.
* Treatment with tyrosine kinase inhibitors or other antileukemic agents or treatments (including HSCT) for longer than 2 weeks, with the exception of HU and/or anagrelide
* Previously documented T315I mutations;
* Uncontrolled congestive heart failure or hypertension;
* Myocardial infarction or unstable angina pectoris within past 12 months;
* Significant arrhythmias, including history or presence of clinically significant ventricular or atrial tachyarrhythmias, clinically significant bradycardias, long QT syndrome and/or QTc > 450 msec on screening ECG (using the QTcF formula). Patients with complete LBBB;
* History of confirmed acute or chronic pancreatitis;
* Other concurrent uncontrolled medical conditions (e.g. uncontrolled diabetes, active or uncontrolled infections, acute or chronic liver and renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol;
* Impaired gastrointestinal function or GI disease that may alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting and diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery);
* Patients with another primary malignancy that is currently clinically significant or requires active intervention;
* Concomitant medications with potential QT prolongation (See link for complete list: http://www.torsades.org/medical-pros/drug-lists/printable-drug-list.cfm);
* Concomitant medications known to interact with CYP450 isoenzymes (CYP 3A4, CYP2C9, CYP2C8, (See link for complete list (http://medicine.iupui.edu/flockhart/table.htm);
* History of significant congenital or acquired bleeding disorder unrelated to cancer;
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy;
* Patients who are pregnant or breastfeeding or adults of reproductive potential not employing an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of nilotinib). Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the entire study and up to 3 months following discontinuation of study drug;
* Treatment with any hematopoietic colony-stimulating growth factors (e.g. G-CSF, GM-CSF) 1 week prior to starting study drug;
* Treatment with other investigational agents (defined as not used in accordance with the approved indication) within 30 days of Day 1;
* Patients unwilling or unable to comply with the protocol.

Note:

Patients who did not meet one or more inclusion or exclusion criteria may be re-screened for this study at a later time if the medical condition is transient and has been appropriately treated (provided they enter the study within 3 months of diagnosis). Date of diagnosis is defined as date of confirmatory bone marrow cytogenetic analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability profile of nilotinib in newly diagnosed CML-AP | 12 month
  The toxicity criteria will be evaluated according to National Cancer Institute - Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 3.0.
To test the efficacy of nilotinib 400 mg BID | 12 months
  To test the efficacy of nilotinib 400 mg BID in inducing complete cytogenetic response (CCyR) at 12 months in newly diagnosed CML-AP patients

SECONDARY OUTCOMES:
Evaluate the rate of complete hematologic response (CHR) | 3 months
  Evaluate the rate of complete hematologic response (CHR) with nilotinib 400 mg BID at 3 months.
Evaluate the Quality of Life | 3, 6, 9, 12, 15, 18 and 24 months
  Evaluate the Quality of Life by FACT-Leu Version 4 questionnaire at 3, 6, 9, 12, 15, 18 and 24 months.
Evaluate the median time to achieve molecular response | uring the first 2 years of treatment
  Evaluate the median time to achieve molecular response and the cumulative probability of obtaining molecular response during the first 2 years of treatment. This will be undertaken through the analysis of the best molecular response at 3, 6, 12, 18 and 24 months. MMR will be preferred and it will be defined as a BCR-ABL/ABL ratio ≤ 0.1% IS using RQ-PCR, but any log reduction between 1 and 4,5 logs will be considered a molecular response.
Evaluate the proportion of patients achieving CCyR | 3, 6, 12, 18 and 24 months or undetectable BCR-ABL levels at 12, 18 and 24 months
  Evaluate the proportion of patients achieving CCyR at 3, 6, 12, 18 and 24 months or undetectable BCR-ABL levels at 12, 18 and 24 months as well as the duration of sustained response.
To correlate the probability of reaching MMR, CMR and CCyR | 2 years
  To correlate the probability of reaching MMR, CMR and CCyR with the risk of progression to blastic phase, relapse and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Biociências SA - Brazil, Study Director — Novartis
Locations (17):
- Brazil (17):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Cuiaba, Mato Grosso do Sul
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Porto Alegre-RS
  - Novartis Investigative Site, Niterói, Rio de Janeiro
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, Santos, São Paulo
  - Novartis Investigative Site, São José, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo